CLINICAL TRIAL: NCT00970229
Title: Evaluation of [123I]MNI-420 and SPECT as a Marker of the Adenosine A2a Receptor in Subjects With Parkinson Disease, Huntington Disease, and Healthy Controls
Brief Title: Evaluation of [123I]MNI-420 and SPECT as a Marker of the Adenosine A2a Receptor in PD, HD and Healthy Subjects.
Acronym: MNI-420
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, David Russell, MD, PhD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-420-01
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson Disease; Huntington Disease
MeSH Terms: conditions — Parkinson Disease; Huntington Disease | interventions — 7-(2-(4-(2-fluoro-4-iodophenyl)piperazin-1-yl)ethyl)-2-(furan-2-yl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidin-5-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [123I]MNI-420 and SPECT Imaging (Experimental): To assess [123I]MNI-420 and SPECT Imaging in PD, HD subjects and similarly aged healthy subjects.
  Interventions: Drug: [123I]MNI-420

INTERVENTIONS:
Drug: [123I]MNI-420 — Subjects will be injected with 8mCi, not to exceed 8.8 mCi (not > 10% of 8 mCi limit)of [123I]MNI-420, followed by SPECT imaging.

SUMMARY:
The underlying goal of this study is to assess [123I]MNI-420 SPECT imaging as a tool to detect A2aR density in the brain of PD and HD research participants to be compared with similarly aged healthy subjects.

DETAILED DESCRIPTION:
* To assess the dynamic uptake and washout of [123I]MNI-420 in brain using single photon emission computed tomography (SPECT) in Parkinson's disease (PD), Huntington's disease (HD), and similarly aged healthy subjects as a potential imaging biomarker of adenosine receptor type A2a (A2aR) in brain
* To acquire initial safety data following injection of [123I]MNI-420

ELIGIBILITY:
Inclusion Criteria:

* Parkinson Subject Selection. Subjects who have a clinical diagnosis of PD will be recruited for this study. The following criteria will be met for inclusion of PD subjects in this study:

  * The participant is 30 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Parkinson disease based on UK Brain Bank Criteria
  * For females, non-child bearing potential or negative urine pregnancy test on day of [123I]MNI-420 injection.
* Huntington Disease Subject Selection. Subjects with a diagnosis of HD will be recruited for this study. The following criteria will be met for inclusion of HD subjects in this study:

  * The participant is 18 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of symptomatic Huntington disease with genetic confirmation
  * Subject is able to provide informed consent as judged by the investigator, or assent can be obtained from the subject and informed consent provided by the appropriate legal representative or next of kin.
  * For females of child-bearing potential, a negative urine pregnancy test on day of [123I]MNI-420 injection.
* Healthy Control Subject Selection. Healthy control subjects who have no neurological disease will be recruited for this study. The following criteria will be met for inclusion of healthy control subjects in this study:

  * The participant is 18 years or older.
  * Written informed consent is obtained.
  * Negative history of neurological or psychiatric illness based on evaluation by a research physician.
  * For females, non-child bearing potential or negative urine or blood pregnancy test on day of [123I]MNI-420 injection.

Exclusion Criteria:

* Parkinson subjects will be excluded from participation for the following reasons:

  * The subject has clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including significant gastrointestinal surgery).
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Clinically significant evidence of vascular disease or alternative neurologic disorder
  * Pregnancy
* Huntington disease subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
  * The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including significant gastrointestinal surgery).
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy
  * Clinically significant evidence of vascular disease or alternative neurologic disorder
* Healthy control subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
  * The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including significant gastrointestinal surgery).
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy
  * Clinically significant evidence of vascular disease or neurologic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-07; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To evaluate [123I]MNI-420 as a quantitative imaging outcome measure of A2aR activity in PD, HD, and healthy subjects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States